CLINICAL TRIAL: NCT06739252
Title: Perioperative Treatment of High-risk Resectable Cholangiocarcinoma With Hepatic Arterial Infusion Chemotherapy (HAIC) Combined With Atezo/Bevacizumab: a Multicenter Phase II Study (NeoBrave CCA)
Brief Title: Perioperative Treatment of High-risk Resectable CCA With HAIC Plus A+T: Neobrave CCA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty of participants enrollment
Sponsor: Peking University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Neobrave-CCA
Record Dates: First submitted 2024-12-01; First posted 2024-12-18 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Intrahepatic Cholangiocarcinoma (Icc); Perihilar Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma; Cirrhosis, Familial, with Pulmonary Hypertension; Klatskin Tumor | interventions — gemcitabine-oxaliplatin regimen; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neobrave (Experimental): Perioperative treatment
  Interventions: Combination Product: Gemcitabine Oxaliplatin and 5FU

INTERVENTIONS:
Combination Product: Gemcitabine Oxaliplatin and 5FU — The perioperative treatment plan includes neoadjuvant therapy and adjuvant therapy. Neoadjuvant therapy consists of three cycles of HAIC combined with atezolizumab and bevacizumab (atezo/bev), while adjuvant therapy includes two cycles of HAIC combined with atezolizumab and bevacizumab (atezo/bev), along with additional capecitabine or tegafur as auxiliary maintenance treatment for three cycles. The total treatment duration for the perioperative period is six months. HAIC regimen: gemcitabine (1,000 mg/m2, 2h, d1) + oxaliplatin (35 mg/m2, 2h, d1-2) + 5-FU (0.75g/m2, 22h, d1-2); atezolizumab (PD-L1 inhibitor): 1200 mg, intravenous infusion, administered within 24 hours before HAIC treatment; bevacizumab: 7.5 mg/kg, intravenously infused before HAIC treatment (bevacizumab use is paused during the third neoadjuvant treatment). Each cycle lasts for three weeks.

SUMMARY:
Among resectable biliary tract cancers (BTC) patients, surgery has historically been the standard treatment, but even with curative surgery, the cure rates remain relatively low, with most patients relapsing in the short term and a 5-year survival rate of approximately 50% or lower.

In BTC, numerous exploratory studies on neoadjuvant treatment have been conducted, yielding varying results, but overall indicating that neoadjuvant therapy can enhance R0 resection rates and prolong survival in certain patients, particularly those with borderline resectable and locally advanced BTC.

Currently, there remains a lack of large prospective randomized controlled phase III clinical trials confirming the exact benefits of neoadjuvant and adjuvant therapies for BTC. The SWOG 1815 study is a randomized, open-label phase III trial comparing GAP with Gemcitabine/Cisplatin (GC) in patients with advanced BTC. In exploratory subgroup analyses, GAP improved mOS compared to GC in patients with locally advanced disease (19.2 vs. 13.7 months; HR 0.67, 95% CI 0.42-1.06, p = 0.09). Thus, patients with locally advanced disease may benefit more from GAP treatment. In another multi-institutional, single-arm, phase II trial, patients received a total of 4 cycles of preoperative GAP (Gemcitabine 800 mg/m2, Cisplatin 25 mg/m2, nab-Paclitaxel 100 mg/m2, administered on days 1 and 8 of a 21-day cycle) before attempting radical surgical resection. The median follow-up time for all patients was 17 months; the disease control rate was 90%. Therefore, the preoperative neoadjuvant therapy of Gemcitabine, Cisplatin, and nab-Paclitaxel for iCCA is feasible and safe, with no adverse effects on perioperative outcomes. More recently, neoadjuvant D + GemCis was confirmed to result in a higher surgical resection rate among patients with locally advanced BTC, and surgical resection was associated with higher survival rates.

The investigators previously explored a prospective phase II study and showed promising results of HAIC using oxaliplatin and 5-fluorouracil for perihilar cholangiocarcinoma (pCCA), with an objective response rate (ORR) of 67.6%, a mPFS of 12.2 months, and a mOS of 20.5 months. Another phase II prospective study enrolled 32 untreated BTC patients and used HAIC combined with anti-PD-1 monoclonal antibody and bevacizumab as a first-line treatment regimen, the ORR was 84.3%, and the disease control rate (DCR) was 96.9%, with one-year PFS and OS rates of 53.8% and 80.4%, respectively.

DETAILED DESCRIPTION:
Biliary tract cancers (BTC), mainly including cholangiocarcinoma and gallbladder cancer, are highly heterogeneous, aggressive malignant tumors with poor prognoses, exhibiting a 5-year survival rate of less than 5%.

About 70% of patients are diagnosed at an advanced localized stage or have distant metastases, losing the chance for surgical cure; among resectable BTC patients, surgery alone has historically been the standard treatment, but even with curative surgery, the cure rates remain relatively low, with most patients relapsing in the short term and a 5-year survival rate of approximately 50% or lower.

The efficacy of neoadjuvant and adjuvant therapies has been validated in other types of cancers and is recommended as standard treatment in various guidelines. In BTC, numerous exploratory studies on neoadjuvant treatment have been conducted, yielding varying results, but overall indicating that neoadjuvant therapy can enhance R0 resection rates and prolong survival in certain patients, particularly those with borderline resectable and locally advanced BTC. With advances in drug research and improvements in treatment protocols, a series of emerging treatment options like combination therapy, targeted therapy, and immunotherapy have significantly improved treatment outcomes, providing favorable conditions for perioperative treatment of BTC.

Currently, there remains a lack of large prospective randomized controlled phase III clinical trials confirming the exact benefits of neoadjuvant and adjuvant therapies for BTC. The SWOG 1815 study is a randomized, open-label phase III trial comparing GAP with Gemcitabine/Cisplatin (GC) in patients with advanced BTC. In exploratory subgroup analyses, GAP improved mOS compared to GC in patients with locally advanced disease (19.2 vs. 13.7 months; HR 0.67, 95% CI 0.42-1.06, p = 0.09); the objective response rate (ORR) for locally advanced disease was 28% vs. 21% (p = 0.74). Thus, patients with locally advanced disease may benefit more from GAP treatment. In another multi-institutional, single-arm, phase II trial including 30 resectable, high-risk iCCA patients (tumor size >5 cm, multiple tumors, major vascular invasion or lymph node involvement seen on imaging), patients received a total of 4 cycles of preoperative GAP (Gemcitabine 800 mg/m2, Cisplatin 25 mg/m2, nab-Paclitaxel 100 mg/m2, administered on days 1 and 8 of a 21-day cycle) before attempting radical surgical resection. The median follow-up time for all patients was 17 months; the disease control rate was 90% (disease progression: 10%, partial response: 23%, stable disease: 67%). Therefore, the preoperative neoadjuvant therapy of Gemcitabine, Cisplatin, and nab-Paclitaxel for iCCA is feasible and safe, with no adverse effects on perioperative outcomes.

With the in-depth research on immune checkpoint inhibitors, during the pre-planned interim analysis of TOPAZ-1 (NCT03875235) (data cutoff date August 11, 2021), the addition of Durvalumab significantly improved OS in patients with advanced BTC compared to the control group receiving GC chemotherapy (hazard ratio [HR], 0.80; 95% confidence interval [CI], 0.66-0.97; p = 0.021). Meanwhile, neoadjuvant D + GemCis was confirmed to result in a higher surgical resection rate among patients with locally advanced BTC, and surgical resection was associated with higher survival rates.

The investigators previously explored a prospective phase II study and showed promising results of HAIC using oxaliplatin and 5-fluorouracil for perihilar cholangiocarcinoma (pCCA), with an objective response rate (ORR) of 67.6%, a mPFS of 12.2 months, and a mOS of 20.5 months. Another phase II single-arm, single-center, prospective study enrolled 32 untreated BTC patients, among which iCCA accounted for 34.4% (11/32), pCCA for 53.1% (17/32), and gallbladder cancer for 12.5% (4/32). Using HAIC combined with anti-PD-1 monoclonal antibody and bevacizumab as a first-line treatment regimen, the ORR was 84.3%, and the disease control rate (DCR) was 96.9%, with one-year PFS and OS rates of 53.8% and 80.4%, respectively.

Based on this study, the investigators plan to conduct a prospective single-arm phase II clinical study to further explore the efficacy and safety of hepatic arterial infusion chemotherapy (HAIC) combined with atezolizumab and bevacizumab (Atezo/Bev) foras perioperative treatment of resectable cholangiocarcinoma with high-risk recurrence factors, while also investigating prognostic and predictive biomarkers related to efficacy to provide new evidence for the perioperative treatment of initially resectable but high-risk recurrence factor intrahepatic and perihilar cholangiocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-80 years, regardless of gender; 2. Diagnosis of intrahepatic cholangiocarcinoma or perihilar cholangiocarcinoma confirmed by pathological tissue/cytological diagnosis; 3. Meeting the criteria for surgical resection; 4. Presence of high-risk recurrence factors: iCCA (single mass >5cm, or multiple lesions, or accompanied by satellite lesions, or accompanied by portal vein/hepatic vein invasion, or CA199 >200U/ml); pCCA (invasion of secondary branches of the bile duct, or invasion of portal vein/hepatic artery, or accompanied by intrahepatic metastasis); 5. Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0-1; 6. Child-Pugh class A; 7. Normal major organ function, meeting the following standards:

1. Blood routine examination:

   A. Hb≥90 g/L; B. ANC≥1.5×10^9/L; C. PLT≥75×10^9/L;
2. Biochemical examination:

A. ALB ≥30g/L; B. ALT and AST<5×ULN; C. TBiL ≤2×ULN; D. Creatinine ≤1.5×ULN; (3) Coagulation function: A. International normalized ratio (INR) ≤1.5×ULN; B. Activated partial thromboplastin time (APTT) ≤1.5×ULN. 8. Subjects voluntarily join this study, sign informed consent, have good compliance, and cooperate with follow-up.

Exclusion Criteria:

1. Regional multiple lymph node metastases or fusion, retroperitoneal lymph node metastases;
2. Peritoneal metastasis, distant metastasis;
3. Previous systemic treatment, including but not limited to chemotherapy, targeted therapy, immunotherapy;
4. Previous local treatment, including but not limited to HAIC, TACE, TARE, ablation, radiotherapy, etc.;
5. Severe hepatic artery variation;
6. Allergy to contrast agents;
7. Allergy to oxaliplatin;
8. Vaccination with live attenuated vaccine within 4 weeks prior to first administration or planned during the study period;
9. Presence of > grade 1 peripheral neuropathy;
10. Presence of any active autoimmune disease or history of autoimmune disease;
11. Complication of other malignancies (except for basal cell or squamous cell skin cancer or cervical carcinoma in situ that was treated curatively);
12. Human immunodeficiency virus (HIV) infection or known acquired immune deficiency syndrome (AIDS);
13. Within 6 months prior to entering the study, occurrences of the following: myocardial infarction, severe/unstable angina, NYHA class II heart failure or above, poorly controlled arrhythmias (including QTcF interval male >450 ms, female >470 ms, QTcF interval calculated using the Fridericia formula), symptomatic congestive heart failure;
14. Hypertension that cannot be well controlled with antihypertensive medications (systolic blood pressure ≥140 mmHg or diastolic pressure ≥90 mmHg);
15. Abnormal coagulation function (INR>1.5 or APTT>1.5×ULN), with bleeding tendency or currently undergoing thrombolytic therapy, anticoagulant therapy, or antiplatelet therapy;
16. Known hereditary or acquired bleeding and thrombosis tendencies, such as hemophilia, coagulation function disorders, thrombocytopenia, splenomegaly, etc.;
17. Significant hemoptysis occurring within 2 months before entering the study, or daily sputum blood volume reaching half a teaspoon (2.5 ml) or more;
18. Patients at risk of gastrointestinal bleeding, including:

(1) Presence of active peptic ulcer lesions; (2) History of melena or hematemesis within the past 3 months; (3) For stool occult blood (+) or (+/-), need to retest stool routine within 1 week; if still (+) or (+/-), esophagogastroduodenoscopy is needed; if ulcers or bleeding diseases are present and considered to have potential bleeding risks by the treating physician; 19. Thrombotic events occurring within 6 months prior to entering the study, such as cerebrovascular accidents (including transient ischemic attacks, intracerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism; 20. Infections requiring drug intervention occurring within 4 weeks prior to first medication (such as requiring intravenous antibiotics, antifungal or antiviral medications), or fever of unknown origin >38.5°C during screening/ prior to first medication; 21. Participation in any other drug clinical trials within 4 weeks prior to first administration; 22. Known history of substance abuse or drug addiction; 23. Presence of other serious physical or mental diseases or abnormal laboratory tests that may increase the risk of participation in the study or interfere with study results, and patients deemed unsuitable for participation in this study by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2024-12-31 (Actual); Primary Completion 2025-12-22 (Actual); Study Completion 2025-12-22 (Actual)

PRIMARY OUTCOMES:
MPR | From the date of treatment beginning to the date of pathological results after the surgery, assessed up to 6 months since the date of treatment beginning
  the proportion of residual active tumor cells ≤50%

SECONDARY OUTCOMES:
pCR | From the date of treatment beginning to the date of pathological results after the surgery, assessed up to 6 months since the date of treatment beginning
  pathological complete response
ORR | Evaluation of tumor burden based on RECIST 1.1 criteria through study completion, an average of once per 3 months.
  objective response rate
DCR | Evaluation of tumor burden based on RECIST 1.1 criteria through study completion, an average of once per 3 months.
  disease control rate
R0 resection rate | From the date of treatment beginning to the date of pathological results after the surgery, assessed up to 6 months since the date of treatment beginning
RFS | From date of treatment beginning until the date of first documented recurrence, assessed up to 100 months
  recurrence-free survival
1-year RFS rate | From enrollment to the date after 1 year of the surgery
OS | From date of treatment beginning until the date of death from any cause, assessed up to 100 months
  overall survival
Number of patients with treatment-related adverse events | Through study completion, an average of once per 1 month.
  Number of patients with AE, treatment-related AE (TRAE), serious adverse event (SAE) assessed by CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaodong Wang, M.D., Study Director — Peking University Cancer Hospital & Institute
Locations (1):
- Peing University Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang X, Hu J, Cao G, Zhu X, Cui Y, Ji X, Li X, Yang R, Chen H, Xu H, Liu P, Li J, Li J, Hao C, Xing B, Shen L. Phase II Study of Hepatic Arterial Infusion Chemotherapy with Oxaliplatin and 5-Fluorouracil for Advanced Perihilar Cholangiocarcinoma. Radiology. 2017 May;283(2):580-589. doi: 10.1148/radiol.2016160572. Epub 2016 Nov 7. PMID 27820684
- [Background] Franssen S, Holster JJ, Jolissaint JS, Nooijen LE, Cercek A, D'Angelica MI, Homs MYV, Wei AC, Balachandran VP, Drebin JA, Harding JJ, Kemeny NE, Kingham TP, Klumpen HJ, Mostert B, Swijnenburg RJ, Soares KC, Jarnagin WR, Groot Koerkamp B. Gemcitabine with Cisplatin Versus Hepatic Arterial Infusion Pump Chemotherapy for Liver-Confined Unresectable Intrahepatic Cholangiocarcinoma. Ann Surg Oncol. 2024 Jan;31(1):115-124. doi: 10.1245/s10434-023-14409-z. Epub 2023 Oct 9. PMID 37814188
- [Background] Franssen S, Soares KC, Jolissaint JS, Tsilimigras DI, Buettner S, Alexandrescu S, Marques H, Lamelas J, Aldrighetti L, Gamblin TC, Maithel SK, Pulitano C, Margonis GA, Weiss MJ, Bauer TW, Shen F, Poultsides GA, Marsh JW, Cercek A, Kemeny N, Kingham TP, D'Angelica M, Pawlik TM, Jarnagin WR, Koerkamp BG. Comparison of Hepatic Arterial Infusion Pump Chemotherapy vs Resection for Patients With Multifocal Intrahepatic Cholangiocarcinoma. JAMA Surg. 2022 Jul 1;157(7):590-596. doi: 10.1001/jamasurg.2022.1298. PMID 35544131
- [Background] Finn RS, Qin S, Ikeda M, Galle PR, Ducreux M, Kim TY, Kudo M, Breder V, Merle P, Kaseb AO, Li D, Verret W, Xu DZ, Hernandez S, Liu J, Huang C, Mulla S, Wang Y, Lim HY, Zhu AX, Cheng AL; IMbrave150 Investigators. Atezolizumab plus Bevacizumab in Unresectable Hepatocellular Carcinoma. N Engl J Med. 2020 May 14;382(20):1894-1905. doi: 10.1056/NEJMoa1915745. PMID 32402160
- [Background] Hack SP, Verret W, Mulla S, Liu B, Wang Y, Macarulla T, Ren Z, El-Khoueiry AB, Zhu AX. IMbrave 151: a randomized phase II trial of atezolizumab combined with bevacizumab and chemotherapy in patients with advanced biliary tract cancer. Ther Adv Med Oncol. 2021 Jul 31;13:17588359211036544. doi: 10.1177/17588359211036544. eCollection 2021. PMID 34377158
- [Background] Hack SP, Zhu AX, Wang Y. Augmenting Anticancer Immunity Through Combined Targeting of Angiogenic and PD-1/PD-L1 Pathways: Challenges and Opportunities. Front Immunol. 2020 Nov 5;11:598877. doi: 10.3389/fimmu.2020.598877. eCollection 2020. PMID 33250900
- [Background] Maithel SK, Keilson JM, Cao HST, Rupji M, Mahipal A, Lin BS, Javle MM, Cleary SP, Akce M, Switchenko JM, Rocha FG. NEO-GAP: A Single-Arm, Phase II Feasibility Trial of Neoadjuvant Gemcitabine, Cisplatin, and Nab-Paclitaxel for Resectable, High-Risk Intrahepatic Cholangiocarcinoma. Ann Surg Oncol. 2023 Oct;30(11):6558-6566. doi: 10.1245/s10434-023-13809-5. Epub 2023 Jun 27. PMID 37368098
- [Background] Utuama O, Permuth JB, Dagne G, Sanchez-Anguiano A, Alman A, Kumar A, Denbo J, Kim R, Fleming JB, Anaya DA. Neoadjuvant Chemotherapy for Intrahepatic Cholangiocarcinoma: A Propensity Score Survival Analysis Supporting Use in Patients with High-Risk Disease. Ann Surg Oncol. 2021 Apr;28(4):1939-1949. doi: 10.1245/s10434-020-09478-3. Epub 2021 Jan 7. PMID 33415559
- [Background] Fruscione M, Pickens RC, Baker EH, Martinie JB, Iannitti DA, Hwang JJ, Vrochides D. Conversion therapy for intrahepatic cholangiocarcinoma and tumor downsizing to increase resection rates: A systematic review. Curr Probl Cancer. 2021 Feb;45(1):100614. doi: 10.1016/j.currproblcancer.2020.100614. Epub 2020 Jun 20. PMID 32622478
- [Background] Patel SP, Othus M, Chen Y, Wright GP Jr, Yost KJ, Hyngstrom JR, Hu-Lieskovan S, Lao CD, Fecher LA, Truong TG, Eisenstein JL, Chandra S, Sosman JA, Kendra KL, Wu RC, Devoe CE, Deutsch GB, Hegde A, Khalil M, Mangla A, Reese AM, Ross MI, Poklepovic AS, Phan GQ, Onitilo AA, Yasar DG, Powers BC, Doolittle GC, In GK, Kokot N, Gibney GT, Atkins MB, Shaheen M, Warneke JA, Ikeguchi A, Najera JE, Chmielowski B, Crompton JG, Floyd JD, Hsueh E, Margolin KA, Chow WA, Grossmann KF, Dietrich E, Prieto VG, Lowe MC, Buchbinder EI, Kirkwood JM, Korde L, Moon J, Sharon E, Sondak VK, Ribas A. Neoadjuvant-Adjuvant or Adjuvant-Only Pembrolizumab in Advanced Melanoma. N Engl J Med. 2023 Mar 2;388(9):813-823. doi: 10.1056/NEJMoa2211437. PMID 36856617
- [Background] Schmid P, Cortes J, Dent R, Pusztai L, McArthur H, Kummel S, Bergh J, Denkert C, Park YH, Hui R, Harbeck N, Takahashi M, Untch M, Fasching PA, Cardoso F, Andersen J, Patt D, Danso M, Ferreira M, Mouret-Reynier MA, Im SA, Ahn JH, Gion M, Baron-Hay S, Boileau JF, Ding Y, Tryfonidis K, Aktan G, Karantza V, O'Shaughnessy J; KEYNOTE-522 Investigators. Event-free Survival with Pembrolizumab in Early Triple-Negative Breast Cancer. N Engl J Med. 2022 Feb 10;386(6):556-567. doi: 10.1056/NEJMoa2112651. PMID 35139274
- [Background] Janssen QP, O'Reilly EM, van Eijck CHJ, Groot Koerkamp B. Neoadjuvant Treatment in Patients With Resectable and Borderline Resectable Pancreatic Cancer. Front Oncol. 2020 Jan 31;10:41. doi: 10.3389/fonc.2020.00041. eCollection 2020. PMID 32083002
- [Background] Franke AJ, Parekh H, Starr JS, Tan SA, Iqbal A, George TJ Jr. Total Neoadjuvant Therapy: A Shifting Paradigm in Locally Advanced Rectal Cancer Management. Clin Colorectal Cancer. 2018 Mar;17(1):1-12. doi: 10.1016/j.clcc.2017.06.008. Epub 2017 Jun 27. PMID 28803718
- [Background] Charfare H, Limongelli S, Purushotham AD. Neoadjuvant chemotherapy in breast cancer. Br J Surg. 2005 Jan;92(1):14-23. doi: 10.1002/bjs.4840. PMID 15635596
- [Background] Burotto M, Wilkerson J, Stein WD, Bates SE, Fojo T. Adjuvant and neoadjuvant cancer therapies: A historical review and a rational approach to understand outcomes. Semin Oncol. 2019 Feb;46(1):83-99. doi: 10.1053/j.seminoncol.2019.01.002. Epub 2019 Jan 26. PMID 30738604
- [Background] Sakamoto Y, Kokudo N, Matsuyama Y, Sakamoto M, Izumi N, Kadoya M, Kaneko S, Ku Y, Kudo M, Takayama T, Nakashima O; Liver Cancer Study Group of Japan. Proposal of a new staging system for intrahepatic cholangiocarcinoma: Analysis of surgical patients from a nationwide survey of the Liver Cancer Study Group of Japan. Cancer. 2016 Jan 1;122(1):61-70. doi: 10.1002/cncr.29686. Epub 2015 Oct 2. PMID 26430782
- [Background] Ishihara S, Horiguchi A, Miyakawa S, Endo I, Miyazaki M, Takada T. Biliary tract cancer registry in Japan from 2008 to 2013. J Hepatobiliary Pancreat Sci. 2016 Mar;23(3):149-57. doi: 10.1002/jhbp.314. Epub 2016 Jan 26. PMID 26699688
- [Background] Wu X, Li M, Wu W, Wang X, Li H, Bao R, Shu Y, Shen J, Gu J, Wang X, Gong W, Peng S, Liu Y. Hepatopancreatoduodenectomy for advanced biliary malignancies. Chin Med J (Engl). 2022 Dec 5;135(23):2851-2858. doi: 10.1097/CM9.0000000000002067. PMID 35916551
- [Background] Valle JW, Lamarca A, Goyal L, Barriuso J, Zhu AX. New Horizons for Precision Medicine in Biliary Tract Cancers. Cancer Discov. 2017 Sep;7(9):943-962. doi: 10.1158/2159-8290.CD-17-0245. Epub 2017 Aug 17. PMID 28818953
- [Background] Kelley RK, Bridgewater J, Gores GJ, Zhu AX. Systemic therapies for intrahepatic cholangiocarcinoma. J Hepatol. 2020 Feb;72(2):353-363. doi: 10.1016/j.jhep.2019.10.009. PMID 31954497
- [Background] Mizrahi JD, Shroff RT. New Treatment Options for Advanced Biliary Tract Cancer. Curr Treat Options Oncol. 2020 Jun 29;21(8):63. doi: 10.1007/s11864-020-00767-3. PMID 32602010
- [Background] Witjes CD, Karim-Kos HE, Visser O, de Vries E, IJzermans JN, de Man RA, Coebergh JW, Verhoef C. Intrahepatic cholangiocarcinoma in a low endemic area: rising incidence and improved survival. HPB (Oxford). 2012 Nov;14(11):777-81. doi: 10.1111/j.1477-2574.2012.00536.x. Epub 2012 Aug 17. PMID 23043667
- [Background] Shaib YH, Davila JA, McGlynn K, El-Serag HB. Rising incidence of intrahepatic cholangiocarcinoma in the United States: a true increase? J Hepatol. 2004 Mar;40(3):472-7. doi: 10.1016/j.jhep.2003.11.030. PMID 15123362
- [Background] Li Y, Yang B, Miao H, Liu L, Wang Z, Jiang C, Yang Y, Qiu S, Li X, Geng Y, Zhang Y, Liu Y. Nicotinamide N -methyltransferase promotes M2 macrophage polarization by IL6 and MDSC conversion by GM-CSF in gallbladder carcinoma. Hepatology. 2023 Nov 1;78(5):1352-1367. doi: 10.1097/HEP.0000000000000028. Epub 2023 Jan 13. PMID 36633260
- [Background] Geng Y, Chen S, Yang Y, Miao H, Li X, Li G, Ma J, Zhang T, Ren T, Li Y, Li L, Liu L, Yang J, Wang Z, Zou L, Liu K, Li Y, Yan S, Cui X, Sun X, Yang B, Zhang L, Han X, Wang C, Chen B, Yue X, Liang W, Ren J, Jia J, Gu J, Li Z, Zhao T, Wang P, Wei D, Qiu S, Xiang D, Xu X, Chen W, He M, Yang L, Wang H, Chen T, Hua R, Wang X, Wu X, Gong W, Wang G, Li M, Zhang W, Shao R, Wu W, Liu Y. Long-term exposure to genistein inhibits the proliferation of gallbladder cancer by downregulating the MCM complex. Sci Bull (Beijing). 2022 Apr 30;67(8):813-824. doi: 10.1016/j.scib.2022.01.011. Epub 2022 Jan 17. PMID 36546234
- [Background] Forner A, Vidili G, Rengo M, Bujanda L, Ponz-Sarvise M, Lamarca A. Clinical presentation, diagnosis and staging of cholangiocarcinoma. Liver Int. 2019 May;39 Suppl 1:98-107. doi: 10.1111/liv.14086. Epub 2019 Mar 25. PMID 30831002
- [Background] Saha SK, Zhu AX, Fuchs CS, Brooks GA. Forty-Year Trends in Cholangiocarcinoma Incidence in the U.S.: Intrahepatic Disease on the Rise. Oncologist. 2016 May;21(5):594-9. doi: 10.1634/theoncologist.2015-0446. Epub 2016 Mar 21. PMID 27000463
- [Background] Razumilava N, Gores GJ. Cholangiocarcinoma. Lancet. 2014 Jun 21;383(9935):2168-79. doi: 10.1016/S0140-6736(13)61903-0. Epub 2014 Feb 26. PMID 24581682
- [Background] Nara S, Esaki M, Ban D, Takamoto T, Shimada K, Ioka T, Okusaka T, Ishii H, Furuse J. Adjuvant and neoadjuvant therapy for biliary tract cancer: a review of clinical trials. Jpn J Clin Oncol. 2020 Dec 16;50(12):1353-1363. doi: 10.1093/jjco/hyaa170. PMID 33037430
- [Background] Kelley RK, Bardeesy N. Biliary Tract Cancers: Finding Better Ways to Lump and Split. J Clin Oncol. 2015 Aug 20;33(24):2588-90. doi: 10.1200/JCO.2015.61.6953. Epub 2015 Jul 20. No abstract available. PMID 26195717